CLINICAL TRIAL: NCT02849171
Title: Pilot Study of 11C-Choline (11C-CH) PET in Assessing Post-treatment True Tumor Progression From Pseudo-progression in High-grade Gliomas
Brief Title: Assessing 11C-Choline (11C-CH) PET to Distinguish True Tumor Progression From Pseudoprogression in High-grade Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-676
Record Dates: First submitted 2016-07-12; First posted 2016-07-29 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-05

CONDITIONS: Brain Cancer
Keywords: 11C-Choline (11C-CH) PET; 16-676; High-grade Gliomas
MeSH Terms: conditions — Brain Neoplasms | interventions — Positron-Emission Tomography; methyl carbon-11 choline

ARMS (1):
- high-grade glioma (Experimental): Eligible patients must have undergone standard radiation (typically 60Gy in 30 fractions), with or without concurrent drug therapy, and have MRI findings consistent with tumor progression and/or pseudoprogression within 24 weeks after completion of radiation. Eligible patients will undergo an 11C-CH PET study within 2 weeks of the standard of care MRI that shows changes concerning for tumor progression vs. pseudoprogression. All patients will then be followed with surveillance brain MRI with and without contrast as per standard of care for a period of 11 months, to assess further progression or stabilization of the lesion. Initial MRI changes are considered to represent pseudoprogression/treatment related changes if the lesion stabilizes or becomes smaller without a change in tumor-related therapy. Otherwise, it will be considered a recurrence should there be progessive radiographic changes.
  Interventions: Device: PET scan; Radiation: C-Choline

INTERVENTIONS:
Device: PET scan
Radiation: C-Choline

SUMMARY:
This is a pilot study. The purpose of this study is to test if an imaging tracer, not approved by the FDA, called 11C-Choline (11C-CH) is useful for evaluating your type of cancer. This tracer is used to perform PET scans. The researchers want to see if the 11C-CH PET scan, using the study tracer 11C-CH, can improve upon the usual scans at diagnosing or monitoring your type of cancer.

In patients with high-grade gliomas, changes on standard MRI of the brain may reflect true tumor growth or inflammatory changes in response to treatment, called pseudo-progression. It is important to distinguish true tumor growth from inflammation since inflammation indicates the tumor is responding to treatment. With standard MRI, it is difficult to determine if changes following treatment are due to tumor growth or inflammation early on. Researchers hope to learn if the investigational tracer, 11C-CH, will be able to distinguish true tumor growth from inflammation more accurately than standard MRI or 18F-FDG PET scans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient is able to provide written informed consent prior to study registration
* Histologically-confirmed high-grade glioma
* Completion of treatment with standard radiation (with or without concurrent therapy).
* Standard gadolinium-enhanced MRI changes that are considered indeterminate for tumor progression vs. treatment-related changes by the neuroradiologist or clinician within 24 weeks of completion of radiation.

Exclusion Criteria:

* Inability to undergo or cooperate with an MRI or PET scan (e.g., claustrophobia, metal implant)
* Renal insufficiency with recent (<3 month old) creatinine > 2.0 mg/dL
* Pregnant or nursing female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07; Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Blasberg, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants have the same disease type, so they were assigned to a single study cohort
Groups:
- High-grade Glioma: Eligible patients must have undergone standard radiation (typically 60Gy in 30 fractions), with or without concurrent drug therapy, and have MRI findings consistent with tumor progression and/or pseudoprogression within 24 weeks after completion of radiation. Eligible patients will undergo an 11C-CH PET study within 2 weeks of the standard of care MRI that shows changes concerning for tumor progression vs. pseudoprogression. All patients will then be followed with surveillance brain MRI with and without contrast as per standard of care for a period of 11 months, to assess further progression or stabilization of the lesion. Initial MRI changes are considered to represent pseudoprogression/treatment related changes if the lesion stabilizes or becomes smaller without a change in tumor-related therapy. Otherwise, it will be considered a recurrence should there be progessive radiographic changes.
  PET scan
  C-Choline
Period: Overall Study
Arm/Group | High-grade Glioma
Started | 8
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Groups:
- High-grade Glioma: All participants have the same disease type, so they were assigned to a single study cohort
Arm/Group | High-grade Glioma
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 58 [44 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: SUV Measures
Description: from 11C-CH PET with evolving changes on brain MRI in high-grade glioma after radiotherapy. In a small subgroup of patients required surgery, tissue will be analyzed for histopathologic correlate. The data gathered will not be considered definitive, but rather will be used to as preliminary data in support of a larger, definitive study.
Time Frame: 1 year
Population: N/A - Data were not collected
Arm/Group | High-grade Glioma
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | High-grade Glioma
All-Cause Mortality (participants affected / at risk) | 7/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-grade Glioma (N=8)
Hyperglycemia (Metabolism and nutrition disorders) | 6
Lymphocyte count decreased (Investigations) | 5
Anemia (Blood and lymphatic system disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 4
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Neutrophil count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT02849171/Prot_SAP_000.pdf